CLINICAL TRIAL: NCT01437826
Title: Evaluation of the Efficacy of a Combination of Micronutrients (Vitamin A, C, E, Selenium and Zinc) in Reducing the Incidence of Colorectal Metachronous Adenomas. A Double Blind, Phase III, Randomized, Placebo-controlled Trial
Brief Title: Antioxidant Supplement and Reduction of Metachronous Adenomas of the Large Bowel: a Double Blind Randomized Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 50% of eligible patients refused to enter the study
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Collaborators: LILT (Italian league against cancer) (Unknown)
Responsible Party: Principal Investigator, Luigina Bonelli, MD, responsible of the unit of secondary prevention and screening, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IST-1988
Record Dates: First submitted 2011-09-14; First posted 2011-09-21 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Colorectal Adenomas
Keywords: chemoprevention; colorectal cancer; metachronous adenoma; randomized trial
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- antioxidants (Experimental): tablets composed of 200 mcg selenium [as l-selenomethionine], 30 mg zinc, 2 mg vitamin A [retinol], 180 mg vitamin C [ascorbic acid] and 30 mg vitamin E [D-α-tocopherol acetate]
  Interventions: Drug: antioxidants
- Sugar pill (Placebo Comparator): placebo had an identical appearance as intervention
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: antioxidants — tablets composed of 200 mcg selenium [as l-selenomethionine], 30 mg zinc, 2 mg vitamin A [retinol], 180 mg vitamin C [ascorbic acid] and 30 mg vitamin E [D-α-tocopherol acetate]
  Other Names: Bio-selenium, Pharma Nord (DK)
  Arms: antioxidants
Drug: placebo — placebo had an identical appearance as intervention
  Other Names: placebo was provided by Pharma Nord
  Arms: Sugar pill

SUMMARY:
The trial was aimed at evaluating the efficacy of a multiagent antioxidant compound (vitamin A, C, E, selenium and zinc) in reducing the incidence of metachronous adenomas of the large bowel after endoscopic polypectomy. This is a randomized study: a 50% reduction in the incidence of metachronous adenomas was expected in patients allocated to the "active" compound (intervention) arm as compared to those assigned to a placebo.

DETAILED DESCRIPTION:
Adenomatous polyps (or adenoma) are benign lesions of the large bowel that are frequent in people aged 60 or more: about one in four of them has at least one adenoma. In time, adenoma could progress to cancer. Even though only a small rate of adenomas will develop into cancer almost 70-80% of colorectal cancer origin from an adenoma and colorectal cancer is one of the most frequent malignant tumors in the western world. Several epidemiological studies showed that subjects who had low intake and/or low blood levels of selenium were at increased risk of developing colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* age 25-75 years
* at least one histologically confirmed adenoma endoscopically removed from the large bowel resulting in a polyp-free colon-rectum (clean colon).

Exclusion Criteria:

* polypectomy performed more than 6 months before enrolment in the trial
* history of Familial Adenomatous Polyposis
* inflammatory bowel disease
* adenoma with invasive carcinoma
* ten or more adenomas
* large sessile adenoma (3 cm or more
* colorectal resection
* invasive cancer at any site
* life-threatening and/or chronic heart, liver or kidney diseases
* current use of vitamin or calcium supplements
* mental disability

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 1988-03; Primary Completion 1996-06 (Actual); Study Completion 1996-06 (Actual)

PRIMARY OUTCOMES:
occurrence of metachronous adenomas or cancer detected during endoscopic follow up examinations | five years

CONTACTS AND LOCATIONS:
Overall Officials: Luigina A Bonelli, MD, Principal Investigator — IRCCS Azienda Ospedale Università San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genova - Italy
Locations (1):
- IRCCS Azienda Ospedale Università San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genova, Italy